CLINICAL TRIAL: NCT00003274
Title: A Randomized Phase II Trial of a Vaccine Combining Tyrosinase /gp100 Peptides Emulsified With Montanide ISA 51 Alone or With a Block Co-Polymer CRL 1005 or With GM-CSF for Patients With Resected Stages IIA and IIB Melanoma Grant Application Title: MART-1/gp100 Immune Responses to a Melanoma Vaccine
Brief Title: Vaccine Therapy in Treating Patients With Stage II Melanoma That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066176 (10M-97-1); LAC-USC-10M971; LAC-USC-FDR001101; NCI-T97-0100
Record Dates: First submitted 1999-11-01; First posted 2004-03-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. It is not yet known what preparation of vaccine therapy is most effective for treating melanoma.

PURPOSE: Randomized phase II trial to study the effectiveness of tyrosinase/gp100 peptide vaccine in treating patients who have stage II melanoma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine immune reactivity in HLA-A2 positive patients with resectable stage IIA or IIB melanoma treated with vaccine comprising tyrosinase peptide and gp100 antigen emulsified in Montanide ISA-51 (ISA-51) alone or in combination with sargramostim (GM-CSF).

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage (IIA vs IIB). Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive vaccine comprising tyrosinase peptide and gp100 antigen emulsified in Montanide ISA-51 (ISA-51) alone subcutaneously (SQ) once a week on weeks 0, 2, 4, 6, 10, 14, 18, and 26. Arm II: Patients receive treatment as in arm I followed by sargramostim (GM-CSF) SQ for 5 days after each vaccination. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients (25 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IIA or stage IIB resectable cutaneous melanoma rendered disease free Clinically uninvolved lymph nodes by physical examination OR Pathologically uninvolved lymph nodes or sentinel lymph nodes after either complete node dissection or selective lymphadenectomy, respectively No evidence of metastatic disease within 28 days prior to definitive surgery HLA-A2 positive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Hematopoietic: No coagulation disorders No significant hematologic abnormality Hepatic: Bilirubin no greater than 2.0 mg/dL No significant liver abnormality Renal: Creatinine no greater than 2.0 mg/dL No significant kidney abnormality Cardiovascular: No major medical illness of the cardiovascular system Pulmonary: No major medical illness of the respiratory system Other: No known allergic reaction to Montanide ISA-51 or sargramostim (GM-CSF) No major systemic infections Not pregnant or nursing HIV negative Hepatitis B surface antigen negative Hepatitis C antibody negative No prior uveitis or autoimmune inflammatory eye disease No active autoimmune disease No other malignancy within past 5 years

PRIOR CONCURRENT THERAPY: At least 1 month since prior adjuvant therapy or any other therapy for cancer Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent steroid therapy Radiotherapy: At least 1 month since prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-03; Primary Completion 2001-09 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan